CLINICAL TRIAL: NCT07397013
Title: Adjustment Technique for Occlusal Stabilizing Splint Used in Temporomandibular Disorders. A Clinical Guide
Brief Title: Adjustment Technique for Occlusal Stabilizing Splint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mai Ahmed Haggag, Assistant Professor, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.26.01.97
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myogenic Temporomandibular Joint Disorders; Internal Derangement of the Tempromandibular Joint; Temporomandibular Disorders (TMDs); Temporomandibular Joint Disc Displacement
Keywords: TMDs; Myogenic Pain; Intraarticular Pain; Disc Displacement; Stabilizing Splint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilizing Splint (3-point of Contact) (Experimental): Stabilizing Splints were adjusted only in centric relation with at least 3-point of contact
  Interventions: Device: Stabilizing Splint(3-point of Contact)
- Stabilizing Splint (Centric and Eccentric) (Experimental): Stabilizing Splints were adjusted in centric relation and in all eccentric movements
  Interventions: Device: Stabilizing Splint (Centric and Eccentric)

INTERVENTIONS:
Device: Stabilizing Splint(3-point of Contact) — These devices are also known as flat plane, inter-occlusal splint, or myo relaxation splint, and are used not only to stabilize the TMJ but also protect the teeth, relax masser etand temporalis muscles, increase inter-discal space, allow the balance of bite forces, and decrease bruxism activity.
  Arms: Stabilizing Splint (3-point of Contact)
Device: Stabilizing Splint (Centric and Eccentric) — Stabilizing Splint (Centric and Eccentric)
  Arms: Stabilizing Splint (Centric and Eccentric)

SUMMARY:
This study aims to clarify the technique of occlusal stabilizing splint adjustment then to assess the overall clinical outcomes and patient satisfaction.

DETAILED DESCRIPTION:
It is reasonable to highlight the occlusal stabilizing splint adjustment protocol as it is important to achieve TMDs' sign and symptom relief. Therefore, the objective of this study is to explain in detail how to adjust the occlusal stabilizing splint properly, as we found few studies that clarify the exact adjustment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the orofacial region (either arthrogenous and/or myogenous) in the last 3 months, who never underwent any type of treatment for TMD's.
* Patients with TMJ internal derangement.
* Age ≥16 years.

Exclusion Criteria:

* Edentulous patients.
* Patients with any systemic disease that could cause joint and/or muscle changes.
* Patients who undergo drug treatment for the condition.
* Current pregnancy or breastfeeding.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Overall Patient Satisfaction | 6 months after using the stabilizing splint
  Using PSPSQ Questionnaire (The patient satisfaction questionnaire comprised three questions assessed using 10-point Likert Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No